CLINICAL TRIAL: NCT07058805
Title: COMPORT: Compartmentalization in Postoperative Radiotherapy for Head and Neck Squamous Cell Carcinoma - A Phase II Clinical Trial
Brief Title: Compartmentalized Postoperative Radiotherapy in Head and Neck Cancer
Acronym: COMPORT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Olgun Elicin (Other)
Collaborators: Clinical Trials Unit, Bern, Switzerland (Unknown); Fond'action contre le cancer (Unknown); University Hospital, Zürich (Other); University Hospital, Basel, Switzerland (Other); Kantonsspital Aarau (Other); Oncology Institute of Southern Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Olgun Elicin, Prof. Dr. med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-BE-2025-01420
Record Dates: First submitted 2025-06-22; First posted 2025-07-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; radiotherapy; Postoperative Radiotherapy; De-escalation; Compartmentalization; Phase II; Quality of life; Bayesian Analysis; TAME; EORTC QLQ-C30; EORTC QLQ-HN43; adjuvant treatment
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Bayesian single-arm phase II design evaluating compartmentalized postoperative radiotherapy in head and neck squamous cell carcinoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compartmentalized postoperative radiotherapy PORT with other without systemic treatment (Experimental): Single-arm study evaluating personalized, pathology- and imaging-guided compartmentalized postoperative radiotherapy (PORT), with or without systemic treatment, in patients with head and neck squamous cell carcinoma. PORT itself or selected target volumes may be omitted based on a predefined algorithm.
  Interventions: Radiation: Compartmentalized Postoperative Radiotherapy

INTERVENTIONS:
Radiation: Compartmentalized Postoperative Radiotherapy — Pathology- and imaging-guided compartmentalized postoperative radiotherapy (PORT), with or without concurrent systemic treatment. Based on a predefined algorithm, PORT or specific anatomical volumes may be omitted. Dose prescription and volumes are risk-adapted.
  Other Names: postoperative adjuvant treatment

SUMMARY:
COMPORT is a multicenter phase II clinical trial evaluating a personalized approach to postoperative radiotherapy in patients with head and neck squamous cell carcinoma (HNSCC). The study investigates whether a risk-adapted, compartmentalized radiotherapy strategy can safely reduce the treatment volume, and thus the side effects, without increasing the risk of tumor recurrence. Eligible patients are those with surgically treated cancers of the oral cavity, oropharynx, larynx, or hypopharynx who have a standard indication for postoperative radiotherapy. The primary outcome is the rate of recurrence in anatomical compartments that would normally be irradiated but are intentionally omitted in this study. COMPORT aims to generate high-level evidence to support a more personalized and less toxic standard of care in postoperative head and neck cancer management.

DETAILED DESCRIPTION:
Background and Rationale:

Head and neck squamous cell carcinoma (HNSCC) is commonly treated with surgery followed by radiotherapy, but conventional large-volume irradiation leads to considerable toxicity. Previous studies, including retrospective work by the COMPORT team (Riggenbach et al. 2024), have shown that a compartmentalized, de-intensified radiotherapy approach may reduce morbidity without compromising oncologic outcomes.

Study Objective:

To evaluate the safety of omitting radiotherapy in selected anatomical compartments that would normally be treated based on standard guidelines (Evans et al. 2018/2025), using a pathology-driven stratification algorithm.

Design:

Bayesian, multicenter, single-arm phase II trial with 50 patients. The primary endpoint is the rate of recurrence in omitted (non-irradiated) compartments within 30 months. Secondary endpoints include loco-regional control, progression-free survival, overall survival, CTCAE-based toxicity scoring (TAME), and patient-reported quality of life (EORTC C30 + HN43).

Analysis Strategy:

The primary analysis will estimate the posterior probability that the recurrence rate in omitted (non-irradiated) compartments remains below a predefined threshold of 18%. If this probability exceeds 90%, the de-escalation strategy will be deemed successful. This would support the rationale for a future phase III randomized trial using a more conservative non-inferiority margin. A predefined interim safety analysis will be conducted once 20 patients have completed at least 6 months of follow-up.

Duration:

Accrual over 24 months, each patient followed for 30 months. Total study period: ~5.5 years.

ELIGIBILITY:
Inclusion criteria

1. ECOG performance status 0-2 at the time of registration
2. ≥18 years of age
3. Baseline assessments and documentation of toxicity using CTCAE v.5 and QoL using EORTC C30 and HN43 questionnaires.
4. Histopathologically confirmed, surgically treated squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx
5. No previous neoadjuvant systemic therapy or previous neoadjuvant systemic therapy (chemotherapy, immunotherapy or combinations) is permitted only if its neoadjuvant use for locally advanced HNSCC is approved by Swissmedic and routinely reimbursed at the time it was administered or if it was administered as part of routine institutional treatment decisions, outside of a clinical trial or other investigational framework.
6. Standard indication for PORT via external beam radiotherapy (with or without concomitant systemic treatment) defined by a multidisciplinary head and neck tumor board (MDT).
7. History and physical examination by treating radiation oncologist within 28 days prior to registration.
8. MRI of the head and neck (or computerized tomography as substitute) with i.v. contrast, if not contraindicated. CT of the chest with i.v. contrast, if not contraindicated. 18FDG-PET/CT can be used instead of CT of the chest. The baseline imaging examinations include the preoperative diagnostic phase and do not have to be repeated if performed within 60 days prior to the enrollment.
9. The multidisciplinary team (MDT) must determine that the patient can safely undergo the standard treatment, which may include PORT with or without additional systemic treatment.
10. Post-menopausal women, or women of child-bearing potential who use or agree to use effective contraception, are not pregnant and agree not to become pregnant during and within 30 days after PORT. A negative pregnancy test before inclusion (within 28 days) into the trial is required for all women with child-bearing potential. Men agree not to father a child during and within three months after PORT.
11. Written informed consent, signed by the patient and the investigator.

Exclusion criteria

1. Synchronous or previous malignancies. Exceptions are curatively treated basal cell carcinoma or SCC of the skin, or in situ carcinoma of the cervix uteri, low- or intermediate- risk prostate cancer, or breast with a progression-free follow-up time of at least 3 years without any remaining disease burden, or other previous malignancy with a progression-free interval of at least 5 years without any remaining active/progressive disease burden regardless whether the treatment is completed or ongoing as a maintenance treatment (e.g. androgen deprivation therapy for prostate cancer).
2. Presence of distant metastases c/pM1.
3. Neoadjuvant systemic therapy administered under a clinical trial protocol or as part of any structured investigational framework not considered standard institutional practice at the time of administration.
4. Previous radiation dose applied to the anatomical sites overlapping with the standard PORT target volumes which may have a potential impact on the delivered dose and/or toxicity profile of the standard PORT.
5. R2 resection of the primary tumor or any involved lymph node.
6. Last oncologic surgery for the index HNSCC performed more than 6 weeks ago.
7. Inadequate reporting of the pathology not conformal with COMPORT algorithm and no possibility of an adequate post-hoc acquisition of the necessary information (see the section 8)
8. Co-existing disease prejudicing survival (expected survival less than 6 months).
9. Active bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
10. Illness expected to preclude PORT within 7 days of registration.
11. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
12. Ongoing participation in another interventional clinical trial which are not exempted by the sponsor. Exceptions may apply depending on the trial methodology (Please contact sponsor for clarification).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate in Omitted Compartments | 30 months from first patient enrollment
  Occurrence of loco-regional recurrence within compartments intentionally omitted from postoperative radiotherapy based on the compartmentalization algorithm compared to the international guidelines (Evans et al. 2018 and 2025).

SECONDARY OUTCOMES:
Loco-regional Control (LRC) | 30 months
  Time to loco-regional failure, including recurrences within irradiated and non-irradiated compartments.
Progression-free Survival (PFS) | 30 months
  Time from registration to disease progression or death from any cause.
Overall Survival (OS) | 30 months
  Time from registration to death from any cause.
Acute and Late Toxicity | 30 months
  Frequency and severity of adverse events using CTCAE v5.0, scored prospectively using the TAME method.
Patient-Reported Global Quality of Life (EORTC QLQ-C30) | 30 months
  The European Organisation for Research and Treatment of Cancer Quality of Life Core Questionnaire-30 (EORTC QLQ-C30) will be used to assess overall and functional quality of life at baseline, post-treatment, and follow-up. The instrument consists of 30 items grouped into multi-item functional scales (Physical, Role, Emotional, Cognitive, Social), symptom scales (e.g., Fatigue, Pain, Nausea/Vomiting), and a global quality of life scale. Each score is linearly transformed to a scale from 0 to 100 according to the official scoring manual. For functional and global health/QoL scales, higher scores represent better functioning or quality of life. For symptom scales, higher scores represent greater symptom burden. The EORTC QLQ-C30 does not generate a total summary score.
Patient-Reported Head and Neck Cancer-specific Quality of Life (EORTC QLQ-HN43) | 30 months
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Cancer module (EORTC QLQ-HN43) will be used to assess specific symptom domains related to head and neck cancer and its treatment. It consists of 43 items grouped into symptom scales and single items (e.g., speech, swallowing, dry mouth, sticky saliva, pain, body image). Each score is linearly transformed to a scale from 0 to 100. Higher scores indicate greater symptom burden. There is no total score. This module is validated for use in conjunction with the EORTC QLQ-C30 in patients with head and neck cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Nannen, Study Director — Inselspital, Bern University Hospital and University of Bern

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing is under consideration but has not yet been finalized. An anonymized individual participant data (IPD) set may be made available upon reasonable request following publication of the primary results and approval by the sponsor and ethics committee.